CLINICAL TRIAL: NCT00322803
Title: International, Multicenter, Randomized, Double-Blind, Placebo Controlled, Two-Period, Cross-Over Study to Demonstrate Safety, Tolerability and Anxiolytic Effects of 600 mg ELB139 Given Orally t.i.d. to Patients With Concurrent Panic Disorder, Challenged by Inhalation of 35% CO2 After a Single Dose and One Week of Treatment
Brief Title: ELB139 Given Orally to Patients With Concurrent Panic Disorder, Challenged by CO2 Inhalation After a Single Dose and One Week of Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: elbion AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ELB139202-05; EudraCT Number:2005-005708-17
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Panic Disorder
Keywords: panic disorder; proof of concept
MeSH Terms: conditions — Panic Disorder | interventions — 1-(4-chlorophenyl)-4-piperidin-1-yl-1,5-dihydroimidazol-2-one

INTERVENTIONS:
Drug: ELB139

SUMMARY:
This study is designed to investigate if 600 mg ELB139 given orally t.i.d. to patients suffering from panic disorder is effective in reducing anxiety evoked by inhalation of 35% CO2 measured by a visual analogue scale after the first intake and after approximately one week of treatment as compared to placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of concurrent panic disorder
* At least 2 panic attacks within the 4 weeks before the screening visit
* Naïve to the CO2 challenge test
* Age 18-65 years (inclusive)
* Ability to comply with all procedures mandated by the study protocol
* Negative pregnancy test and adequate contraceptive measures

Exclusion Criteria:

* History of poly-pharmacotherapy for panic disorder or treatment resistance
* Any current psychiatric Axis I DSM-IV diagnosis other than panic disorder, except concurrent simple phobia
* History of abuse of benzodiazepines or tolerance to effects of benzodiazepine
* Any concomitant psychotropic medication
* Evidence of impaired hepatic, renal or cardiac functions
* Participation in any drug trial in the preceding 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-05; Study Completion 2006-10

PRIMARY OUTCOMES:
degree of subjective anxiety as measured on a Visual Analogue Scale for Anxiety(VAS-A) assessed immediately after the CO2-challenge (VAS-A-post)
difference of the degree of anxiety measured as the difference between the pre- and post challenge scores on the Visual Analogue Scale for Anxiety (VAS-A-delta)

SECONDARY OUTCOMES:
Total Symptom Score assessed immediately after CO2 challenge (TSS-post)
Difference of the Total Symptoms Score (TSS) measured as the difference between the pre- and post challenge scores (TSS-delta)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Griez, Prof Dr, Principal Investigator — Academic Anxiety Center and Department of Psychiatry & Neuropsychology; Maastricht University
Locations (3):
- Germany (2):
  - Charité - University Clinics Berlin, Berlin
  - Emovis, The institute of emotional health, Berlin
- Academic Anxiety Center and Department of Psychiatry & Neuropsychology; Maastricht University, Maastricht, Netherlands